CLINICAL TRIAL: NCT01977456
Title: Phase 2 The Combined Approach to Lysis Utilizing Eptifibatide and Rt-PA in Acute Ischemic Stroke-Full Dose Regimen(CLEAR-FDR)
Brief Title: Study of the Combination Therapy of Rt-PA and Eptifibatide to Treat Acute Ischemic Stroke (CLEAR-FDR)
Acronym: CLEAR-FDR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arthur Pancioli (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Arthur Pancioli, sub investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P50NS044283-13 (NIH); P50NS044283-13 (NIH)
Record Dates: First submitted 2013-10-18; First posted 2013-11-06 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-10

CONDITIONS: Stroke; Brain Infarction
Keywords: acute ischemic stroke; stroke; rt-PA, thrombolytic; t-PA; recombinant tissue plasminogen activator; Activase; eptifibatide; Integrilin; fibrinolytic agents; clot dissolving; blood clot
MeSH Terms: conditions — Stroke; Brain Infarction; Ischemic Stroke; Thrombosis | interventions — Eptifibatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eptifibatide (Experimental): All subjects will receive the standard dose of IV rt-PA. All subjects will promptly receive an IV bolus of 135mcg/kg eptifibatide followed by an IV infusion of 0.75 mcg/kg/min eptifibatide for 2 hours.
  Interventions: Drug: Eptifibatide

INTERVENTIONS:
Drug: Eptifibatide — IV Eptifibatide is an approved drug by the Food and Drug Administration as a treatment for blood clots causing heart attack and chest pain.Eptifibatide inhibits platelet aggregation by blocking activated platelets from binding fibrinogen.
  Other Names: Integrilin

SUMMARY:
The primary goal of this trial is to determine if individuals with acute ischemic stroke treated with a full dose of IV recombinant tissue plasminogen activator (rt-PA) plus IV eptifibatide started within 3 hours of symptom onset are more likely to have a better outcome than individuals treated with standard IV rt-PA alone.

DETAILED DESCRIPTION:
The Combined Approach to Lysis Utilizing Eptifibatide and rt-PA in Acute Ischemic Stroke-Full Dose Regimen (CLEAR-FDR Stroke Trial) is a Phase II trial and part of the Specialized Program on Translational Research in Acute Stroke (SPOTRIAS). The overall goals of SPOTRIAS are to enhance delivery of acute stroke patient care and train acute stroke translational researchers.

Stroke most often occurs when blood flow to the brain stops because it is blocked by a blood clot. When a blood clot blocks the blood supply to the brain, parts of the brain may not get enough blood and oxygen to survive. As a result, permanent brain damage can occur, which can affect a person's ability to walk, talk, and function independently. In order to reduce the risk of permanent damage, it is important to restore blood flow to the brain as quickly as possible.

rt-PA, used alone, is already approved by the Food and Drug Administration (FDA) as treatment for patients with a stroke caused by blockage of an artery in the brain and when given within 3 hours of the onset of stroke symptoms. Eptifibatide is also already FDA-approved as a treatment for blood clots causing heart attack. The investigational aspect of this study is the use of eptifibatide for a stroke victim in combination with rt-PA.

The CLEAR Stroke Trial demonstrated that the combination of low dose rt-PA plus eptifibatide can be safely given to acute ischemic stroke patients within 3 hours of symptom onset.

The CLEAR-ER Stroke Trial demonstrated that the combination of medium dose rt-PA plus eptifibatide can be safely given to acute ischemic stroke patients within 3 hours of symptom onset.

The CLEAR-FDR Stroke Trial is designed to provide data concerning the risks when combining eptifibatide with full dose intravenous rt-PA in 30 acute ischemic stroke patients within 3 hours of symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a serious measurable neurological deficit on the NIH Stroke Scale due to focal brain ischemia.
* An NIH Stroke Scale score >5 at the time the rt-PA is begun.
* Age: 18 through 85 years (i.e. candidates must have had their 18th birthday, but not had their 86th birthday).
* Intravenous rt-PA therapy must be initiated within 3 hours of onset of stroke symptoms.

Exclusion Criteria:

* History of stroke in the past 3 months.
* Previous intra-cranial hemorrhage, neoplasm, subarachnoid hemorrhage, or arterial venous malformation.
* Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT scan is normal.
* Hypertension at time of treatment; systolic BP > 185 or diastolic > 110 mmHg or aggressive measures to lower blood pressure to below these limits are needed.
* Presumed septic embolus.
* Presumed pericarditis including pericarditis after acute myocardial infarction.
* Recent (within 30 days) surgery or biopsy of parenchymal organ.
* Recent (within 30 days) trauma, with internal injuries or ulcerative wounds.
* Recent (within 90 days) severe head trauma or head trauma with loss of consciousness.
* Any active or recent (within 30 days) serious systemic hemorrhage.
* Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency; or oral anticoagulant therapy with International Normalized Ratio (INR) > 1.7.
* Baseline lab values: positive urine pregnancy test, glucose < 50 or > 400 mg/dl, platelets <100,000 /mm3, Hct <25 %, or creatinine > 4 mg/dl.
* Ongoing renal dialysis, regardless of creatinine.
* Subjects who received Low Molecular Weight heparins (such as Dalteparin, Enoxaparin, Tinzaparin) as deep vein thrombosis (DVT) prophylaxis or in full dose within the previous 24 hours.
* Subjects who received heparin or a direct thrombin inhibitor (such as bivalirudin, argatroban, or lepirudin) within 48 hours from screening must have had a normal partial prothrombin time (PTT).
* Subjects who received Factor Xa inhibitors (such as fondaparinux) or direct thrombin inhibitors (such as dabigatran) within the last 4 days.
* Arterial puncture at a non-compressible site or a lumbar puncture in the previous 7 days.
* Seizure at onset of stroke.
* Pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations.
* Other serious, advanced, or terminal illness or any other condition that the investigator feels would pose a significant hazard to the patient if rt-PA or eptifibatide therapy were initiated.
* Patients whose peripheral venous access is so poor that they are unable to have two standard peripheral intravenous lines started.
* Current participation in another research drug treatment protocol. Patient cannot start another experimental agent until after 90 days.
* Informed consent is not or cannot be obtained.
* Any known history of amyloid angiopathy.
* High density lesion consistent with hemorrhage of any degree.
* Significant mass effect with midline shift.
* Large (more than 1/3 of the middle cerebral artery) regions of clear hypodensity on the baseline CT scan. Sulcal effacement and/or loss of grey-white differentiation alone are not contraindications for treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Opeolu Adeoye, MD, Principal Investigator — University of Cincinnati
Locations (8):
- United States (8):
  - St. Elizabeth Healthcare System Edgewood, Edgewood, Kentucky
  - St. Elizabeth Healthcare Florence, Florence, Kentucky
  - St. Elizabeth Healthcare Ft. Thomas, Fort Thomas, Kentucky
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Jewish Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio

REFERENCES:
- [Result] Adeoye O, Sucharew H, Khoury J, Vagal A, Schmit PA, Ewing I, Levine SR, Demel S, Eckerle B, Katz B, Kleindorfer D, Stettler B, Woo D, Khatri P, Broderick JP, Pancioli AM. Combined Approach to Lysis Utilizing Eptifibatide and Recombinant Tissue-Type Plasminogen Activator in Acute Ischemic Stroke-Full Dose Regimen Stroke Trial. Stroke. 2015 Sep;46(9):2529-33. doi: 10.1161/STROKEAHA.115.010260. Epub 2015 Aug 4. PMID 26243231

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eptifibatide
Started | 27
Completed | 22
Not Completed | 5
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Arm/Group | Eptifibatide
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 27
National Institutes of Health Stroke Scale Score (NIHSS) [Median (Inter-Quartile Range); unit: score] — NIHSS score: A 43 point ordinal scale (0 to 42) measuring severity of stroke. 0 (no measurable effect), 42 (dead)
  score | 12 [9 to 16]

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Who Experience Symptomatic Intracerebral Hemorrhage (sICH).
Description: Any ICH related to a decline in neurologic status or the development of new neurologic symptoms which in the judgment of the clinical investigator was related to the ICH. Judgment of significant neurological decline was made by the local clinical investigator
Time Frame: within 36 hours after stroke onset
Measure: Number; unit: participants
Arm/Group | Eptifibatide
Number analyzed (Participants) | 27
participants | 1

2. Secondary Outcome: The Number of Patients Who Experience Any Intracerebral Hemorrhage (ICH).
Description: Any ICH symptomatic (as defined above) or asymptomatic (that visualized on CT or MRI only)
Time Frame: within 36 hours after stroke onset
Measure: Number; unit: participants
Arm/Group | Eptifibatide
Number analyzed (Participants) | 27
participants | 2

3. Secondary Outcome: The Number of Patients Who Develop Parenchymal Hemorrhage Types 1( PH-1) and 2 (PH-2).
Description: Any parenchymal hemorrhage types PH-1 or PH-2 as visualized on CT
Time Frame: within 36 hours after stroke onset
Measure: Number; unit: participants
Arm/Group | Eptifibatide
Number analyzed (Participants) | 27
participants | 1

4. Other Pre Specified Outcome: The Number of Participants With Good Outcomes According to the Modified Rankin Score.
Description: Modified Rankin score (mRS) dichotomized to good outcome (mRS 0-1 or return to baseline), poor outcome (all others including death). Results reported are good outcome.
Time Frame: 90 days from the date of stroke onset
Measure: Number; unit: participants
Arm/Group | Eptifibatide
Number analyzed (Participants) | 27
participants | 17

ADVERSE EVENTS:
Time Frame: Serious adverse events are monitored through 90 days. Non-serious adverse events are monitored through day 3 or discharge
Arm/Group | Eptifibatide
Serious Adverse Events (participants affected / at risk) | 4/27
Other Adverse Events (participants affected / at risk) | 17/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eptifibatide (N=27)
Anaemias nonhaemolytic and marrow depression (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrhythmias (Cardiac disorders) | 1 (1)
Heart failures (Cardiac disorders) | 1 (1)
Diabetic complications (Endocrine disorders) | 1 (2)
Glucose metabolism disorders (incl diabetes mellitus) (Endocrine disorders) | 1 (1)
General system disorders NEC (General disorders) | 2 (2)
Diabetic complications (Metabolism and nutrition disorders) | 1 (2)
Glucose metabolism disorders (incl diabetes mellitus) (Metabolism and nutrition disorders) | 1 (1)
Neurological disorders NEC (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eptifibatide (N=27)
Coagulopathies and bleeding diatheses (excl thrombocytopenic) (Blood and lymphatic system disorders) | 2 (2)
White blood cell disorders (Blood and lymphatic system disorders) | 2 (2)
Cardiac arrhythmias (Cardiac disorders) | 4 (4)
Gastrointestinal motility and defaecation conditions (Gastrointestinal disorders) | 2 (2)
Gastrointestinal signs and symptoms (Gastrointestinal disorders) | 3 (3)
Infections - pathogen unspecified (Infections and infestations) | 3 (3)
Electrolyte and fluid balance conditions (Metabolism and nutrition disorders) | 2 (2)
Musculoskeletal and connective tissue disorders NEC (Musculoskeletal and connective tissue disorders) | 2 (2)
Neurological disorders NEC (Nervous system disorders) | 2 (2)
Anxiety disorders and symptoms (Psychiatric disorders) | 2 (2)
Genitourinary tract disorders NEC (Renal and urinary disorders) | 3 (3)
Urinary tract signs and symptoms (Renal and urinary disorders) | 2 (2)
Epidermal and dermal conditions (Skin and subcutaneous tissue disorders) | 2 (2)
Skin vascular abnormalities (Skin and subcutaneous tissue disorders) | 2 (2)
Decreased and nonspecific blood pressure disorders and shock (Vascular disorders) | 2 (2)
Vascular haemorrhagic disorders (Vascular disorders) | 7 (8)

LIMITATIONS AND CAVEATS:
Small sample size and open design. Did not include endovascular therapy patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No